CLINICAL TRIAL: NCT04928456
Title: Augmentation of Immune Response to COVID-19 mRNA Vaccination Through Osteopathic Manipulative Treatment Including Lymphatic Pumps
Brief Title: Augmentation of Immune Response to COVID-19 mRNA Vaccination Through OMT With Lymphatic Pumps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: American College of Osteopathic Physicians (Unknown); American Osteopathic Foundation (Unknown); Osteopathic Physicians and Surgeons of California (Unknown); Xavier-Nichols Foundation (Unknown)
Responsible Party: Principal Investigator, Jesus Sanchez, Professor of Family Medicine, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FB21/IRB026
Record Dates: First submitted 2021-06-11; First posted 2021-06-16 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: COVID-19; OMT; Vaccination; Osteopathic manipulation
MeSH Terms: conditions — COVID-19 | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized, no-treatment control group, OMT intervention group with a parallel group design.
Who Masked: Care Provider, Investigator
Masking Description: Care providers will not be involved with any of the data acquisition or analysis. Investigators will be blinded to which participants are in each group and will collect data using only subject numbers provided on labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT Intervention Arm (Experimental): OMT will include:
  1. Myofascial release of the thoracic inlet: gentle pressure applied to shoulders and neck to move the tissue in different directions with a gentle motion.
  2. Pectoral traction: The armpit will be contacted with the finger pads of the doctor and each side will be gently grasped and have a slow pulling force applied towards the shoulders.
  3. Diaphragm release with MFR: The doctor will touch below the ribs on each side and will apply gentle pressure and move the tissue from side to side.
  4. Splenic pump: below the ribs on the left hand-side, the doctor will apply pressure and release pressure several times to create a vibration over the area just below the ribs.
  5. Thoracic pump: The doctor will place their hands over the chest wall on each side and will apply pressure and release pressure several times to generate a pumping action of about 100 times in one minute.
  Treatment will last 5 minutes with each technique lasting 1 minute.
  Interventions: Other: Osteopathic Manipulative Treatment (OMT)
- Control (No Intervention): Participants in the control group will undergo the same assessments as the OMT intervention arm and will receive their vaccinations, but will not receive any OMT.

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment (OMT) — Osteopathic Manipulative Treatment (OMT) involves a number of hands-on techniques that are meant to address somatic dysfunction in the body as a part of the osteopathic approach to treating patients. There will be five techniques in total used in the study treatment plan.
  Arms: OMT Intervention Arm

SUMMARY:
This study will evaluate the effectiveness of utilizing Osteopathic Manipulative Treatment (OMT) procedures as an addition to current mRNA COVID-19 vaccines in terms of enhancing the immune response of participants as assessed by looking for increased levels and duration of antibody titers.

DETAILED DESCRIPTION:
The COVID-19 pandemic has taken many lives, caused millions to become ill, many hospitalized, it has wreaked havoc on our economy, our mental states, and many other aspects of our lives. Vaccines have provided the world with much needed relief against the pandemic but concerns of vaccine escape and naturally waning antibody titers remain in place. The emergence of new strains are a cause of concern. Standard vaccine protocol does not currently utilize the osteopathic medical approach. It has yet to be seen if OMT improves the immune system's response to the COVID-19 spike protein provided by vaccines. Prior research using OMT with lymphatic treatments has shown improved outcomes for hospitalized patients, patients with various diseases, and improved vaccine delivery for Hepatitis B vaccines. This randomized clinical trial will assess the effectiveness of the addition of OMT to COVID-19 vaccination procedures. Individuals will be recruited from those who present at the WesternU vaccine clinic for their first COVID-19 vaccination and from the incoming classes, current classes, faculty, and staff of the 9 colleges at the university. Volunteers will be consented to the study if they qualify and will be randomly assigned to either the control group who will only receive their vaccinations or into the OMT intervention group who will receive OMT provided by an osteopathic physician or an osteopathic OMM Teaching Fellow the day of each of their two vaccinations and the day following the two vaccinations.

Baseline blood samples will be taken for all subjects enrolled in the study. These baseline blood samples will be analyzed for IgG against nucleocapsid as a control to see if there was any previous infection since this would not be present in vaccinated individuals who had never been exposed and contracted COVID-19 and IgG against the spike protein which would help to track the immunity built up in response to the vaccine. Both groups will then receive their first vaccination and only the OMT intervention group will then undergo OMT after receiving their vaccine. The OMT group will return the next day to receive treatments for a second time. Both groups will have blood drawn for IgG vaccine titers against spike protein at 7 days, 21 days, 28 days, 35 days, 3 months, 6 months, and 12 months. Both groups will be asked to report any side effects and any medications used to combat these side effects throughout the entirety of the study. If a subject were to feel symptoms of COVID-19 during the study they would be asked to take a RT-PCR test so that the infection could be verified and tested for the strain type.

OMT modalities that will be used include myofascial release of the thoracic inlet, pectoral traction, diaphragm release with myofascial release, splenic pump, and thoracic pump. All techniques will be performed on the individuals with each technique lasting a total of 1 minute and the entire treatment lasting a total of 5 minutes.

The primary comparison will be the titer of antibodies at each point of each volunteer as expressed as a percentage of the base line pre-vaccination titer between the intervention group (receiving OMT) compared to the control group (not receiving OMT).

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 and 65 years old
* Will be receiving the mRNA COVID-19 vaccine at Western University of Health Sciences
* Have signed an informed consent form
* Have not previously received a COVID-19 vaccine

Exclusion Criteria:

* Have contraindications to vaccine and any significant reactions to vaccines
* Have any primary or secondary immune deficiencies or autoimmune disease/immunocompromised
* Have symptoms of COVID-19 at the time of enrollment (eg. Fever, headaches, muscle pain, sore throat, coughing, loss of smell, loss of taste, etc.)
* Have already received a COVID-19 vaccine
* Are using any immune altering medications such as corticosteroids, cyclospoin, tacrolimus, and pimecrolimus
* Are unable to receive OMT with lymphatic techniques due to open wounds, fractures, anuresis, necrotizing faciitis, congestive heart failure, or unstable cardiac conditions
* Are pregnant or breastfeeding
* Are less than 18 years of age or more than 65 years of age
* Were previously treated for COVID-19 with serum transfer or immunological treatments
* Are on anti-coagulation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
IgM antibody titer levels Percentage Change. | At 1 week, 3 weeks, 4 weeks, 5 weeks, 3 months, 6 months and 1 year post- vaccination.
  Percentage change from baseline in IgM assay levels of pre-vaccination titer vs IgM assay levels in subjects receiving control treatment (no OMT) vs subjects receiving intervention treatment (OMT).
IgG antibody titer levels Percentage Change | At 1 week, 3 weeks, 4 weeks, 5 weeks, 3 months, 6 months and 1 year post- vaccination.
  Percentage change from baseline in IgG assay levels of pre-vaccination titer vs IgG assay levels in subjects receiving control treatment (no OMT) vs subjects receiving intervention treatment (OMT).
IgM and IgG antibody titer duration | At 3 months, 6 months and 1 year post- vaccination.
  Time in days in which levels of IgM and IgG assay remain above detectable levels in subjects receiving control treatment (no OMT) vs subjects receiving intervention treatment (OMT) after vaccination.

SECONDARY OUTCOMES:
Medication Usage | Through study completion, an average of 1 year
  Assessment of medications that subjects used to negate side effects using a medication log.
Adverse Effects/Side Effects | Through study completion, an average of 1 year
  Reported side effects from the vaccines or adverse effects experienced from OMT.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Sanchez, DO, Principal Investigator — Professor of Family Medicine
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No